CLINICAL TRIAL: NCT07276568
Title: A Clinical Study on the Safety and Tolerability of Hepatocyte-like Cells in Patients With Liver Failure and Small-for-Size Syndrome
Brief Title: Safety and Tolerability of Hepatocyte-like Cell Therapy for Liver Failure and Small-for-Size Syndrome
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhi-Jun Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhi-Jun Zhu, Principal Investigator, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFH20251030001
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Acute Liver Failure; Acute on Chronic Liver Failure (ACLF); Chronic Liver Failure; Small-for-size Syndrome
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure; End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acute Liver Failure (Experimental): On the basis of standard medical therapy, patients will receive an intramuscular injection of CiPS-derived hepatocyte cells into the rectus sheath.
  The method, dose, timing, and treatment course of rectus sheath injection of CiPS-derived hepatocyte cells (adjusted by body weight for adults/adolescents) are set as follows:
  ① Cell quantity: A dose-escalation design (ranging from 1.6 × 10⁷/kg to 1.7 × 10⁸/kg) will be adopted. Treatment will initiate at the lower dose (1.6 × 10⁷/kg). Upon successful safety review, the dose will be gradually escalated up to a maximum of 1.7 × 10⁸/kg.
  Interventions: Drug: Hepatocyte-like cell administration via rectus sheath intramuscular injection
- Acute-on-Chronic Liver Failure (Experimental): On the basis of standard medical therapy, patients will receive an intramuscular injection of CiPS-derived hepatocyte cells into the rectus sheath.
  The method, dose, timing, and treatment course of rectus sheath injection of CiPS-derived hepatocyte cells (adjusted by body weight for adults/adolescents) are set as follows:
  ① Cell quantity: A dose-escalation design (ranging from 1.6 × 10⁷/kg to 1.7 × 10⁸/kg) will be adopted. Treatment will initiate at the lower dose (1.6 × 10⁷/kg). Upon successful safety review, the dose will be gradually escalated up to a maximum of 1.7 × 10⁸/kg.
  Interventions: Drug: Hepatocyte-like cell administration via rectus sheath intramuscular injection
- Chronic liver failure (Experimental): On the basis of standard medical therapy, patients will receive an intramuscular injection of CiPS-derived hepatocyte cells into the rectus sheath.
  The method, dose, timing, and treatment course of rectus sheath injection of CiPS-derived hepatocyte cells (adjusted by body weight for adults/adolescents) are set as follows:
  ① Cell quantity: A dose-escalation design (ranging from 1.6 × 10⁷/kg to 1.7 × 10⁸/kg) will be adopted. Treatment will initiate at the lower dose (1.6 × 10⁷/kg). Upon successful safety review, the dose will be gradually escalated up to a maximum of 1.7 × 10⁸/kg.
  Interventions: Drug: Hepatocyte-like cell administration via rectus sheath intramuscular injection
- Small-for-Size Syndrome (Experimental): On the basis of standard medical therapy, patients will receive an intramuscular injection of CiPS-derived hepatocyte cells into the rectus sheath.
  The method, dose, timing, and treatment course of rectus sheath injection of CiPS-derived hepatocyte cells (adjusted by body weight for adults/adolescents) are set as follows:
  ① Cell quantity: A dose-escalation design (ranging from 1.6 × 10⁷/kg to 1.7 × 10⁸/kg) will be adopted. Treatment will initiate at the lower dose (1.6 × 10⁷/kg). Upon successful safety review, the dose will be gradually escalated up to a maximum of 1.7 × 10⁸/kg.
  Interventions: Drug: Hepatocyte-like cell administration via rectus sheath intramuscular injection

INTERVENTIONS:
Drug: Hepatocyte-like cell administration via rectus sheath intramuscular injection — On the basis of standard medical therapy, patients will receive an intramuscular injection of CiPS-derived hepatocyte cells into the rectus sheath.
  The method, dose, timing, and treatment course of rectus sheath injection of CiPS-derived hepatocyte cells (adjusted by body weight for adults/adolescents) are set as follows:
  ① Cell quantity: A dose-escalation design (ranging from 1.6 × 10⁷/kg to 1.7 × 10⁸/kg) will be adopted. Treatment will initiate at the lower dose (1.6 × 10⁷/kg). Upon successful safety review, the dose will be gradually escalated up to a maximum of 1.7 × 10⁸/kg.

SUMMARY:
To evaluate the safety, tolerability, and preliminary efficacy of intramuscular injection of hepatocyte-like cells into the rectus sheath in patients with liver failure (including acute liver failure, acute-on-chronic liver failure, and chronic liver failure) and small-for-size syndrome, with the ultimate goal of improving survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with liver failure or small-for-size syndrome based on clinical presentation.

（Acute Liver Failure (ALF) An acute onset of liver failure characterized by hepatic encephalopathy of grade II or higher within 4 weeks, in a patient without pre-existing liver disease.

Acute-on-Chronic Liver Failure (ACLF) A complex clinical syndrome characterized by acute deterioration of liver function, triggered by precipitating events, in patients with underlying chronic liver disease (with or without cirrhosis). It manifests as single or multiple organ failure(s) and is associated with high short-term mortality (28-day mortality rate ≥ 15%).

Chronic Liver Failure (CLF) A state of chronic hepatic decompensation occurring progressively in patients with cirrhosis. It is primarily characterized by recurrent ascites and/or hepatic encephalopathy resulting from progressively declining liver function.

Small-for-Size Syndrome (SFSS) Diagnosis is established according to the International Liver Transplantation Society (ILTS) 2023 guidelines on SFSS.） ② Patients must agree to undergo intramuscular injection of cells into the rectus sheath.

Exclusion Criteria:

-

Subjects meeting any of the following criteria will be excluded from the study:

1. Presence of severe, life-threatening extrahepatic systemic diseases.
2. Uncontrolled active infection or hemorrhage.
3. Pregnancy or lactation in female patients.
4. History of severe allergic reactions or known hypersensitivity to CiPS-derived cell products or blood products.
5. Inability to undergo phlebotomy due to peripheral vascular collapse.
6. Inability or unwillingness to provide informed consent or comply with the study procedures.
7. Unwillingness to receive CiPS-based therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | 1 year following injection
Adverse Reaction Rate | within 1 year following injection
  Adverse reactions related to hepatocyte-like cell injection can be categorized into two types: i) injection-related adverse reactions (such as bleeding and infection), and ii) cell product-related adverse reactions (including but not limited to immune rejection and tumorigenicity).

SECONDARY OUTCOMES:
Serum Alanine Aminotransferase (ALT) | Blood samples will be collected at before treatment, 8 hours, 12 hours, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  ALT levels in U/L will be measured from blood samples. The outcome will be reported as the change from baseline in ALT levels at each specified time point.
Serum Aspartate Aminotransferase (AST) | Blood samples will be collected at before treatment, 8 hours, 12 hours, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  AST levels in U/L will be measured from blood samples. The outcome will be reported as the change from baseline in AST levels at each specified time point.
Serum Total Bilirubin | Blood samples will be collected at before treatment, 8 hours, 12 hours, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  Total bilirubin levels in mg/dL (or μmol/L) will be measured from blood samples. The outcome will be reported as the change from baseline in total bilirubin levels at each specified time point.
Serum Direct Bilirubin | Blood samples will be collected at before treatment, 8 hours, 12 hours, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  Direct bilirubin levels in mg/dL (or μmol/L) will be measured from blood samples. The outcome will be reported as the change from baseline in direct bilirubin levels at each specified time point.
Plasma Ammonia | Blood samples will be collected at before treatment, 8 hours, 12 hours, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  Ammonia levels in μmol/L will be measured from blood samples. The outcome will be reported as the change from baseline in plasma ammonia levels at each specified time point.
Heart Rate | Measured at before treatment, and at 0.5, 1, 2, 4, 8, 12 hours post-treatment, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  Heart rate will be measured in beats per minute (bpm) in a supine or sitting position after the participant has rested for at least 5 minutes. The outcome will be reported as the change from baseline in heart rate at each specified time point.
Respiratory Rate | Measured at before treatment, and at 0.5, 1, 2, 4, 8, 12 hours post-treatment, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  Respiratory rate will be measured in breaths per minute (brpm). The outcome will be reported as the change from baseline in respiratory rate at each specified time point.
Blood Pressure) | Measured at before treatment, and at 0.5, 1, 2, 4, 8, 12 hours post-treatment, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  Blood pressure will be measured in millimeters of mercury (mmHg) in a supine or sitting position after the participant has rested for at least 5 minutes.
Consciousness Level as assessed by Glasgow Coma Scale (GCS) | Assessed at before treatment, and at 0.5, 1, 2, 4, 8, 12 hours post-treatment, and on days 1, 3, 7, 14, as well as at months 1, 3, 6, and 12 post-treatment.
  The level of consciousness will be assessed using the Glasgow Coma Scale (GCS). The GCS total score ranges from 3 to 15, with a lower score indicating a lower level of consciousness. The outcome will be reported as the absolute GCS score and the change from baseline at each specified time point.
Graft Morphological Stability on T2-weighted Fat-Suppressed (T2W-FS) MRI | MRI assessments will be performed at baseline (post-transplantation), and at Day 28, Month 3, 6, and 12 post-transplantation.
  The graft site within the left rectus abdominis muscle will be assessed by T2W-FS MRI for morphological stability. The outcome is based on the presence or absence of significant changes in location, shape, and size compared to the baseline (post-engraftment) scan. The absence of mass effect, displacement, or deformation of the surrounding muscle will be documented. Stability in these parameters over time will be considered a favorable outcome, while significant deviation will be reported as an adverse event.
Graft Signal Characteristics on T2-weighted Fat-Suppressed (T2W-FS) MRI | MRI assessments will be performed at baseline (post-transplantation), and at Day 28, Month 3, 6, and 12 post-transplantation.
  The graft site will be assessed by T2W-FS MRI for signal intensity characteristics. The outcome is based on the signal intensity and pattern (e.g., homogeneous, stippled, nodular) relative to the surrounding normal muscle tissue. A stable or resolving signal pattern without the development of focal, nodular, or mass-like high signal intensity will be considered a favorable outcome. The development of new or evolving high-signal areas suggestive of abnormal growth will be reported.
Absence of Abnormal Fat Deposition on T1-weighted Fat-Suppressed (T1W-FS) MRI | MRI assessments will be performed at baseline (post-transplantation), and at Day 28, Month 3, 6, and 12 post-transplantation.
  The graft site will be assessed by T1W-FS MRI for the absence of abnormal fat deposition, a key indicator for teratoma formation. The outcome is a binary assessment (Yes/No) of whether the signal intensity of the graft region is isointense to surrounding normal muscle tissue.

IPD SHARING:
Plan to Share IPD: No